CLINICAL TRIAL: NCT05632237
Title: Evaluation of a Family Strengthening Program Evaluation in Sierra Leone to Prevent Family Separation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Christian Alliance for Orphans (Unknown); Helping Children Worldwide (Unknown); Child Reintegration Centre (Unknown)
Responsible Party: Principal Investigator, Sarah Neville, PhD, Boston College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: cafo
Record Dates: First submitted 2022-11-09; First posted 2022-11-30 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-08

CONDITIONS: Parent-Child Relations; Emotion Regulation; Economic Problems; Parenting
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Masking Description: During baseline data collection, participants were not yet assigned to arms, so all parties were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family strengthening program (Experimental)
  Interventions: Behavioral: Family strengthening program
- Care as usual (No Intervention): These participants have already been receiving case management from the Child Reintegration Centre prior to the study, and they will continue to receive care as usual, which is to receive normal case management visits without this added Family Strengthening Program component. Case management consists of a social work staff alternating between visiting children at home or at school each month to provide supervision, coaching, counseling, assessments, and identification of additional support needs.

INTERVENTIONS:
Behavioral: Family strengthening program — Phase I: 2-day Family Strengthening Workshop. The specific topics included in the workshop include: emotions, Body Progressive Muscle Relaxation, body stretch, self care, apologizing, routines to promote attachment, teamwork, saving, delayed gratification, anticipating unexpected expenses, identifying family strengths and values.
  Phase II: Case management with family strengthening curriculum. Curriculum is delivered over the course of four visits (about 3 months), some of which involve both caregiver and child while others are just for the caregiver. Topics included are using appropriate discipline, effective communication for family problem-solving, and home budgeting.
  Arms: Family strengthening program

SUMMARY:
In Sierra Leone, poverty and challenges with family functioning can lead to family separation, and children may go to live on the street or enter residential care institutions/orphanages. Helping Children Worldwide (HCW), a non-profit organization with over 20 years of experience in Sierra Leone, has developed a two-part Family Strengthening Program delivered by their program partners in Sierra Leone, the Child Reintegration Centre, to improve families financial literacy and attachment between caregivers and children, with the ultimate goal of preventing family separation. The hypothesis of this study is that the Family Strengthening Program program is effective at (1) changing parenting behaviors, (2) improving emotional regulation, (3) improving caregiver-child attachment, and (4) improving financial literacy in dyads consisting of children ages 9-13 and their caregivers.

ELIGIBILITY:
Inclusion criteria:

1. Dyads must consist of a principal child (the one whose situation initiated their involvement with the Child Reintegration Centre) and their primary caregiver (as defined by the Child Reintegration Centre as the person in the family primarily responsible for the health and wellbeing of the principal child and is noted as such in their case file)
2. Primary child is ages 9-13
3. Dyad is actively participating in Child Reintegration Centre services (i.e., child must have been seen by the case manager in the last month)
4. Dyad lives in the Bo area.

Exclusion criterion:

(1) Family has been assessed by the Child Reintegration Centre to be in active crisis, i.e., specific concerns about the child being at-risk or unsafe (suspicions of abuse or neglect).

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2022-10-16 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Caregiver and child change in emotional regulation as measured by the Difficulties in Emotional Regulation (DERS) scale | Baseline: Up to 2 months before intervention; Endline: Up to 2 months after intervention
Change in child attachment as measured by the Inventory of Parent and Peer Attachment (IPPA) | Baseline: Up to 2 months before intervention; Endline: Up to 2 months after intervention
Change in caregiver- and child-reported use of punishment by caregiver | Baseline: Up to 2 months before intervention; Endline: Up to 2 months after intervention
  Measures developed for this study tailored for context; e.g., flogging child with hand or cane, public shaming, withholding food
Change in self-reported economic well-being | Baseline: Up to 2 months before intervention; Endline: Up to 2 months after intervention
  Measures developed for this study tailored for context and intervention content; e.g., awareness of income/spending, saving and budgeting behaviors, ability to pay for unexpected expense

SECONDARY OUTCOMES:
Change in child- and caregiver-reported parenting behaviors by caregiver | Baseline: Up to 2 months before intervention; Endline: Up to 2 months after intervention
  Measures developed for this study tailored for context and intervention content; e.g., asking child about their life, spending one-on-one time with child, physically showing affection, giving compliments/praise, using a routine, apologizing, providing emotional support

CONTACTS AND LOCATIONS:
Locations (1):
- the Child Reintegration Centre, Bo, Sierra Leone

IPD SHARING:
Plan to Share IPD: No